CLINICAL TRIAL: NCT04899921
Title: A Blinded, Randomized Phase 2 Study of Troriluzole in Combination With Ipilimumab and Nivolumab in Patients With Melanoma Brain Metastases Previously Treated With Anti-PD-1 Therapy
Brief Title: Troriluzole or Placebo Plus Ipi Plus Nivo in Mel Brain Mets
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to poor enrollment
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Biohaven Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Ann W. Silk, MD MS, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-675
Record Dates: First submitted 2021-04-16; First posted 2021-05-25 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Melanoma; Metastatic Melanoma
Keywords: Melanoma; Metastatic Melanoma; Metastatic Melanoma, Brain
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Nivolumab; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Ipilimumab + Nivolumab + Troriluzole [Phase I dose level 1] (Experimental): Phase I dose level 1 participants received nivolumab 1 mg/kg and ipilimumab 3 mg/kg intravenously (IV) on day 1 of each 21-day cycle and the original starting troriluzole dose of 140 mg orally in the morning as well as 280 mg orally in the evening every day of each 21-day cycle. Participants were treated until disease progression or unacceptable toxicity.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Drug: Troriluzole
- Ipilimumab + Nivolumab + Troriluzole [Phase II] (Experimental): Participants will be randomly assigned and receive:
  12 Week Induction Phase: Nivolumab at pre-determined dose followed by ipilimumab at predetermined dose every 3 weeks, with 21 consecutive days defined as a treatment cycle. Troriluzole self-administered at a predetermined dose orally twice a day
  36 Week Maintenance Phase: Nivolumab will be administered every 4 weeks, with 28 consecutive days defined as a treatment cycle. Troriluzole self administered at a predetermined dose orally twice a day. No ipilimumab will be given in the maintenance phase.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Drug: Troriluzole
- Ipilimumab + Nivolumab + Placebo [Phase II] (Experimental): Participants will be randomly assigned and receive:
  12 Week Induction Phase: Nivolumab at pre-determined dose followed by ipilimumab at predetermined dose every 3 weeks, with 21 consecutive days defined as a treatment cycle. Placebo self-administered at a predetermined dose orally twice a day
  36 Week Maintenance Phase: Nivolumab will be administered every 4 weeks, with 28 consecutive days defined as a treatment cycle. Placebo self administered at a predetermined dose orally twice a day. No ipilimumab will be given in the maintenance phase.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Drug: Placebo
- Ipilimumab + Nivolumab + Troriluzole [Phase I dose level 2] (Experimental): Phase I dose level 2 participants received nivolumab 1 mg/kg and ipilimumab 3 mg/kg intravenously (IV) on day 1 of each 21-day cycle and troriluzole 140 mg twice per day orally. Participants were treated until disease progression or unacceptable toxicity.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Drug: Troriluzole
- Ipilimumab + Nivolumab + Troriluzole [Phase I dose level 3] (Experimental): Phase I dose level 3 participants received nivolumab 1 mg/kg and ipilimumab 3 mg/kg intravenously (IV) on day 1 of each 21-day cycle and troriluzole 140 mg/day orally. Participants were treated until disease progression or unacceptable toxicity.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Drug: Troriluzole

INTERVENTIONS:
Drug: Ipilimumab — Intravenous injection
  Other Names: Yervoy
Drug: Nivolumab — Intravenously (IV) into the vein
  Other Names: Opdivo
Drug: Troriluzole — Taken orally
  Other Names: BHV-4157; Trigriluzole; FC-4157
  Arms: Ipilimumab + Nivolumab + Troriluzole [Phase I dose level 1]; Ipilimumab + Nivolumab + Troriluzole [Phase I dose level 2]; Ipilimumab + Nivolumab + Troriluzole [Phase I dose level 3]; Ipilimumab + Nivolumab + Troriluzole [Phase II]
Drug: Placebo — Taken orally
  Other Names: Sugar Pill
  Arms: Ipilimumab + Nivolumab + Placebo [Phase II]

SUMMARY:
The purpose of this research is to test the safety and effectiveness of the investigational combination of Troriluzole, ipilimumab, and nivolumab, and to learn whether this combination works in treating melanoma that has spread to the brain.

DETAILED DESCRIPTION:
This is a multi-center, double-blind, randomized, phase II signal-detection trial with a non-randomized safety run-in to assess the efficacy and safety of adding troriluzole to ipilimumab/nivolumab induction and nivolumab maintenance in patients with melanoma that has metastasized to the brain. Measuring the shrinking or growth of melanoma in participants will allow researchers to learn about these study drugs and provide information on the safety and effectiveness of this combination in treating melanoma.

The U.S. Food and Drug Administration (FDA) has not approved Troriluzole as a treatment for any disease. The U.S. Food and Drug Administration (FDA) has approved nivolumab, ipilimumab, and the combination of these two drugs as treatment options for melanoma that has metastasized to the brain.

Ipilimumab and nivolumab are drugs that treat cancer by blocking certain molecules in the body. This blocking action prevents other molecules from binding to cells involved in the immune system. With these changes, the immune system is more likely to become active, and will react more intensely when activated. The immune system is able to destroy cancer cells and reduce the size of tumors, so activating the immune system is an important part of cancer treatment. Ipilimumab blocks a molecule called cytotoxic T-lymphocyte-associated protein-4 (CTLA-4), which normally decreases the activation of the immune system by binding to T-Cells, which are important immune system cells that can attack cancer cells. Nivolumab blocks a molecule called programmed death receptor-1 (PD-1), which also normally decreases the activation of the immune system.

Troriluzole is a drug that modulates glutamate, the most abundant excitatory neurotransmitter in the human body. The primary mode of action of Troriluzole is reducing synaptic levels of glutamate. This may change parts of the immune system in the brain, which is could improve treatment outcomes with anti-cancer drugs such as ipilimumab and nivolumab that can work in the brain. This study is testing Troriluzole's ability to increase the effectiveness of ipilimumab and nivolumab treatment in melanoma that has spread to the brain, as well as testing the safety of the combination of these three drugs.

Participation in this research is expected to last up to 4 years: 1 year of treatment and 3 years of follow up.

About 108 subjects will take part in this research.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed melanoma. All melanoma subtypes are included, except for ocular melanoma.
* Participants must have measurable disease in the brain (intraparenchymal brain metastases), defined as at least one lesion that can be accurately measured by magnetic resonance imaging (MRI) in at least one dimension as ≥5 mm and ≤ 3 cm in longest diameter. See Section 11 (Measurement of Effect) for the evaluation of measurable disease. Measurable disease in the extracranial compartment (body) is not required. Measurable lesions may not have received previous treatment with radiation therapy. Prior stereotactic radiation therapy (SRT; e.g. GammaKnife, CyberKnife) is allowed for lesions other than the lesions selected as measurable target lesions. Prior craniotomy with resection of brain metastases is allowed.
* Participants must have received prior systemic treatment with anti-PD-1 therapy (e.g. pembrolizumab, or nivolumab) in any setting (neoadjuvant, adjuvant or metastatic). Prior anti-CTLA-4 monotherapy is allowed (e.g. ipilimumab). Prior targeted therapy (e.g. BRAF inhibitors, MEK inhibitors) is allowed.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of troriluzole in participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* ECOG performance status 0 or 1 (see Appendix A).
* Participants must have adequate organ and marrow function as defined below:

  * absolute neutrophil count ≥1,000/mcL
  * total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN), or in the case of Gilbert's disease ≤ 3x ULN
  * AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* The effects of troriluzole on the developing human fetus are unknown. For this reason and because ipilimumab is a pregnancy category C, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence from heterosexual intercourse) prior to study entry, for the duration of study participation, and 4 months after completion of all study drugs. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of all study drugs.
* Ability to swallow pills.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Ocular subtype of melanoma.
* Cytologically confirmed leptomeningeal metastases, or convincing imaging evidence of leptomeningeal spread.
* Prior whole brain radiation therapy (WBRT).
* Prior combination therapy with concurrent ipilimumab (3 mg/kg IV) + nivolumab (1 mg/kg IV) in the 24 months prior to the date of registration.
* Participants who have had systemic therapy (immunotherapy, chemotherapy, or targeted therapy), radiotherapy, or major surgery within 3 weeks prior to the date of registration.
* Participants who require immediate local treatment (surgical resection or radiosurgery) of brain metastases due to neurological symptoms, or brain metastases located in sensitive areas of the brain requiring immediate local treatment.
* Participants who have required systemic steroids to manage neurologic symptoms (seizures, cerebral edema, severe headache, nausea/vomiting, etc.) within 1 week prior to the date of registration.
* Participants who are receiving any other investigational agents for cancer or neurologic disease.
* Extreme claustrophobia that would interfere with performing brain MRIs or severe allergy to gadolinium contrast.
* History of severe or life-threatening allergic reactions attributed to compounds of similar chemical or biologic composition to troriluzole, riluzuole, ipilimumab, or nivolumab.
* Second primary malignancy that is a competing cause of death in the opinion of the treating investigator (prognosis < 6 months).
* Patients with a history of solid organ transplant, or allogeneic bone marrow transplant.
* Active autoimmune disease or any other condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other systemic immunosuppressive medications within 3 weeks of registration.
* History of grade 4 immune related adverse event from prior cancer treatment, (with the exception of asymptomatic elevation of serum amylase or lipase).
* History of immune-related adverse event from prior cancer immunotherapy treatment that has not improved to grade 0-1 (with the exception of patients with ongoing thyroid, adrenal or gonadal insufficiency requiring continued medical treatment, vitiligo, or asymptomatic elevation of serum amylase or lipase).
* Participants receiving any medications or substances that are inhibitors or inducers of the liver enzyme Cytochrome P-450 CYP1A2, including fluvoxamine, cimetidine, amiodarone, efavirenz, fluoroquinolones (including ciprofloxacin and levofloxacin), fluvoxamine, furafylline, interferon, methoxsalen, mibefradil, or ticlopidine. These medications must be discontinued at least 7 days prior to registration.
* Participants with uncontrolled intercurrent illness.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and nursing (breastfeeding) women are excluded from this study because the effects of troriluzole on the developing human fetus are unknown, and because ipilimumab is pregnancy category

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann W Silk, MD, MS, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Aden D, Sureka N, Zaheer S, Chaurasia JK, Zaheer S. Metabolic Reprogramming in Cancer: Implications for Immunosuppressive Microenvironment. Immunology. 2025 Jan;174(1):30-72. doi: 10.1111/imm.13871. Epub 2024 Oct 27. PMID 39462179

RESULTS

PARTICIPANT FLOW:
Groups:
- Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 2]: Phase I dose level 2 participants received nivolumab 1 mg/kg and ipilimumab 3 mg/kg intravenously (IV) on day 1 of each 21-day cycle and troriluzole 140 mg twice per day orally. Participants were treated until disease progression or unacceptable toxicity,
Period: Overall Study
Arm/Group | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 1] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 2] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 3]
Started | 0 | 0 | 0
Completed (Terminated with 1 patient enrolled, no data due to patient privacy.) | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Terminated with1 patient enrolled; no data due to patient privacy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 1] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 2] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 3] | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical
Age, Continuous [unit: years] — years
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Median Global Progression-Free Survival (PFS)
Description: Global PFS is defined as the time from random assignment to the earlier of death or documented disease progression in the intracranial or extracranial compartments. The follow-up of patients who have neither died nor progressed will be censored at the date of the last follow-up visit. Disease assessment was based on RECIST 1.1 for all extracranial lesions and modified RECIST 1.1 for all brain lesions. Per RECIST 1.1 for target lesions: PD is at least a 20% increase in sum LD, taking as reference the smallest sum on study with at least 5 mm absolute increase. For non-target lesions, progression-free means no new lesions or unequivocal progression on existing non-target lesions or not evaluated,
Time Frame: Participants would be followed up to 5 years.
Population: Terminated with 1 patient enrolled; no data due to patient privacy.
Arm/Group | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 1] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 2] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 3]
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Median Overall Survival (OS)
Description: OS was defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive. Estimates of OS would be from a PHMC model.
Time Frame: Participants were followed up to 5 years.
Population: Terminated with 1 patient enrolled; no data due to patient privacy.
Arm/Group | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 1] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 2] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 3]
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Intracranial Response Rate (RR)
Description: Intracranial response rate was defined as the proportion of participants who have achieved complete response (CR) or partial response (PR) based on modified RECIST 1.1.
Time Frame: From enrollment to end of treatment up to 5 years
Population: Terminated with 1 patient enrolled; no data due to patient privacy.
Arm/Group | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 1] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 2] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 3]
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Intracranial Progression-free Survival (PFS)
Description: Intracranial PFS was defined as the time from first dose of study therapy to documented intracranial progression or death, whichever occurs first. Per modified RECIST 1.1 for target lesions: PD is at least a 20% increase in sum LD, taking as reference the smallest sum on study with at least 5 mm absolute increase. For non-target lesions, progression-free means no new lesions or unequivocal progression on existing non-target lesions or not evaluated.
Time Frame: From date of randomization until the date of first documented intracranial progression or date of death from any cause, whichever came first, assessed up to 5 years.
Population: Terminated with 1 patient enrolled; no data due to patient privacy.
Arm/Group | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 1] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 2] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 3]
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Extracranial Response Rate (RR)
Description: The extracranial response rate was defined as the proportion of participants who have achieved complete response or partial response based on Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) for all extracranial lesions.
Time Frame: From enrollment to end of treatment up to 5 years
Population: Terminated with 1 patient enrolled; no data due to patient privacy.
Arm/Group | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 1] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 2] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 3]
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Extracranial Progression-free Survival (PFS)
Description: Extracranial PFS is defined as the time from first dose of study therapy to documented extracranial progression (per RECIST) or death, whichever occurs first. Evaluated using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1)39 for all extracranial lesions and modified RECIST 1.1 for all brain lesions
Time Frame: From date of randomization until the date of first documented extracranial progression or date of death from any cause, whichever came first, assessed up to 5 years.
Population: Terminated with 1 patient enrolled; no data due to patient privacy.
Arm/Group | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 1] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 2] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 3]
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE Version 5.0
Description: The number and proportion of adverse events, graded as defined by CTCAE version 5.0 will be tabulated by type and grade.
Time Frame: From enrollment to end of treatment up to 5 years
Population: Terminated with 1 patient enrolled; no data due to patient privacy.
Arm/Group | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 1] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 2] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 3]
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Number of Induction
Description: Number of induction cycles was defined as the number of induction cycles administered.
Time Frame: From enrollment to end of treatment up to 5 years
Population: Terminated with 1 patient enrolled; no data due to patient privacy.
Arm/Group | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 1] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 2] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 3]
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Number of Maintenance Cycles
Description: Number of maintenance cycles was defined as the number of maintenance cycles administered.
Time Frame: From enrollment to end of treatment up to 5 years
Population: Terminated with 1 patient enrolled; no data due to patient privacy.
Arm/Group | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 1] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 2] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 3]
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Corticosteroids Usage
Description: Corticosteroids usage was defined by number of participants who require prednisone ≥1 mg/kg or equivalent.
Time Frame: From enrollment to end of treatment up to 5 years
Population: Terminated with 1 patient enrolled; no data due to patient privacy.
Arm/Group | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 1] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 2] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 3]
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Frequency of Clinically-indicated Stereotactic Radiation Therapy to the Brain
Description: Frequency of clinically-indicated stereotactic radiation therapy to the brain was defined as the number of participants who received on-study brain-directed stereotactic radiation.
Time Frame: From enrollment to end of treatment up to 5 years
Population: Terminated with 1 patient enrolled; no data due to patient privacy.
Arm/Group | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 1] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 2] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 3]
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Frequency of Clinically-indicated Surgical Intervention to the Brain
Description: Frequency of clinically-indicated surgical intervention to the brain was defined as the number of participants who received on-study surgical intervention to the brain.
Time Frame: From enrollment to end of treatment up to 5 years
Population: Terminated with 1 patient enrolled; no data due to patient privacy."
Arm/Group | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 1] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 2] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 3]
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Observation period regarding adverse event was up to 5 years from the start of treatment.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv4. All remaining events regardless of treatment attribution were classified as Other AEs. Per the source vocabulary (CTCAEv5.0) there is a category "Other, specify" for each system organ class. No further data is available to specify classification beyond this general term.
Arm/Group | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 1] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 2] | Ipilimumab + Nivolumab + Troriluzole [Phase I Dose Level 3]
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT04899921/Prot_SAP_000.pdf